CLINICAL TRIAL: NCT03742232
Title: A Multicentre Randomized Parallel Group Phase IV Study Comparing the Bowel Cleansing Efficacy, Safety and Tolerability of PLENVU® Versus SELG-ESSE® Using a 2-Day Split Dosing Regimen.
Brief Title: Study Comparing the Bowel Cleansing Efficacy of PLENVU® Versus SELG-ESSE® Using a 2-Day Split Dosing Regimen.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2063
Record Dates: First submitted 2018-11-13; First posted 2018-11-15 (Actual); Last update posted 2020-08-27 (Actual); Status verified 2020-08

CONDITIONS: Colon Polyp; Colon Adenoma; Colon Lesion
MeSH Terms: conditions — Colonic Polyps | interventions — polyethylene glycol 3350; Polyethylene Glycols

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PLENVU (Experimental): PLENVU® supplied as two powder-for-oral-solution formulations. One formulation contains PEG3350, sodium sulphate and electrolytes, and the second formulation contains PEG3350, sodium ascorbate, ascorbic acid, and electrolytes.
  Interventions: Drug: PEG3350
- SELG-ESSE (Active Comparator): SELG-ESSE® supplied as powder-for-oral-solution containing PEG4000, simethicone, sodium sulphate and sodium bicarbonate, and electrolytes.
  Interventions: Drug: Macrogol 4000

INTERVENTIONS:
Drug: PEG3350 — PLENVU® supplied as two powder-for-oral-solution formulations. One formulation contains PEG3350, sodium sulphate and electrolytes, and the second formulation contains PEG3350, sodium ascorbate, ascorbic acid, and electrolytes.
  PLENVU® Administration: 2-Day Split-Dosing Regimen (to commence in the evening of the day before colonoscopy).
  Arms: PLENVU
Drug: Macrogol 4000 — SELG-ESSE® supplied as powder-for-oral-solution containing PEG4000, simethicone, sodium sulphate and sodium bicarbonate, and electrolytes.
  SELG-ESSE® Administration: 2-Day Split-Dosing Regimen (to commence in the evening of the day before colonoscopy).
  Arms: SELG-ESSE

SUMMARY:
This study is a multicentre randomized parallel group phase IV study comparing the bowel cleansing efficacy, safety and tolerability of PLENVU® (a 1 litre PEG Bowel Cleansing Solution) versus SELG-ESSE® (a 4 litre PEG Bowel Cleansing Solution) using a 2-Day Split Dosing Regimen.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must provide written informed consent.
2. Male and female outpatients and inpatients aged: ≥18 to ≤85 years undergoing a screening, surveillance or diagnostic colonoscopy.
3. Females of child-bearing potential must have a negative pregnancy test at Screening and at Visit 2 and must be practising one of the following methods of birth control and agree to continue with the regimen throughout the study period:

   * Oral, implantable, or injectable contraceptives (for a minimum of three months before study entry) in combination with a condom;
   * Intrauterine device in combination with a condom; Double barrier method (condom*, and occlusive cap [diaphragm or cervical/vault caps] with spermicidal foam/gel/film/ cream/suppository); *A female condom and a male condom should not be used together as friction between the two can result in either product failing.

   If any female patient has a positive pregnancy test at Visit 2, they will be excluded from further participation in the study for the efficacy evaluation, i.e. they will not undergo the colonoscopy procedure. The Investigator will be required to arrange a colonoscopy procedure outside of the study.

   Note: The above birth control methods do not apply to females who are postmenopausal or surgically sterile i.e. 12 months of natural (spontaneous) amenorrhea or 6 weeks' post-surgical bilateral oophorectomy with or without hysterectomy or hysterectomy, or whose sole sexual partner has had a vasectomy and has received medical assessment of the surgical success.
4. Willing, able and competent to complete the entire study and to comply with instructions.

Exclusion Criteria:

1. Patients with past history within last 12 months or current episode of severe constipation (requiring repeated use of laxatives/enema or physical intervention before resolution), known or suspected ileus, gastrointestinal obstruction, gastric retention, bowel perforation, toxic colitis or megacolon.
2. Patients with ongoing severe acute Inflammatory Bowel Disease (IBD).
3. Patients who have had previous significant gastrointestinal surgeries, including colonic resection, sub-total colectomy, abdomino-perineal resection, de-functioning colostomy, Hartmann's procedure and defunctioning ileostomy or other similar surgeries involving structure and function of the small or large colon.
4. Regular use of laxatives or colon motility altering drugs (i.e. more than 2-3 times per week) in the last 28 days prior to the Screening Visit and/or laxative use within 72 hours prior to administration of the preparation.
5. Patients with active intestinal bleeding episodes
6. Known glucose-6-phosphate dehydrogenase (G6PD) deficiency.
7. Known phenylketonuria.
8. Known hypersensitivity to polyethylene glycols, ascorbic acid and sulfates (not including sulfa-based products) or any other component of the investigational product or comparator.
9. Past history within the last 12 months or evidence of any on-going clinically relevant electrocardiogram (ECG) abnormalities (e.g. arrhythmias).
10. History of uncontrolled hypertension with systolic blood pressure >170 mmHg and diastolic blood pressure >100 mmHg.
11. Patients with cardiac insufficiency NYHA grades III or IV.
12. Patients with severe renal insufficiency.
13. Patients with known liver disease of grades B and C according to the Child Pugh classification.
14. Patients suffering from dehydration at screening as evaluated by the Investigator from physical examination.
15. Patients with pre-existing clinically significant electrolyte abnormalities, or dehydration.
16. Patients with impaired consciousness that might predispose them to pulmonary aspiration.
17. Patients undergoing colonoscopy for foreign body removal and/or decompression.
18. Patients who are pregnant or lactating, or intending to become pregnant during the study.
19. Clinically relevant findings on physical examination based on the Investigator's judgment.
20. History of drug or alcohol abuse within the 12 months prior to dosing.
21. Concurrent participation in an investigational drug or device study or participation within three months of study entry.
22. Patients who, in the opinion of the Investigator, should not be included in the study for any reason, including inability to follow study procedures, e.g. cognitively impaired, debilitated or fragile patients.
23. Patients who are ordered to live in an institution on court or authority order.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 399 (Actual)
Dates: Start 2018-10-31 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Bowel cleansing efficacy | 1 Day of colonoscopy
  To evaluate the overall bowel cleansing efficacy of 2-day split-dosing with PLENVU compared to a 2-day split-dosing regimen with SELG-ESSE®, graded according to the Boston Bowel Preparation Scale (BBPS) in patients undergoing screening, surveillance or diagnostic colonoscopy.

SECONDARY OUTCOMES:
Polip Detection Rate | 1 Day of colonoscopy
  To assess the overall Polip Detection Rate with PLENVU compared to SELG-ESSE
Adenoma Detection Rate | 1 Day of colonoscopy
  To assess the overall Adenoma Detection Rate with PLENVU compared to SELG-ESSE;
Adverse events | 4 days after colonscopy
  To assess the incidence of adverse events in PLENVU group comparing SELG-ESSE arm

CONTACTS AND LOCATIONS:
Locations (5):
- Italy (5):
  - Centro di Riferimento Oncologico, Aviano, Italia
  - Fondazione Poliambulanza, Brescia, Italia
  - Nuovo Regina Margherita Hospital, Roma, Italia
  - ISMETT, Palermo
  - Humanitas Research Hospital, Rozzano

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Repici A, Spada C, Cannizzaro R, Traina M, Maselli R, Maiero S, Galtieri A, Guarnieri G, Di Leo M, Lorenzetti R, Capogreco A, Spadaccini M, Antonelli G, Zullo A, Amata M, Ferrara E, Correale L, Granata A, Cesaro P, Radaelli F, Minelli Grazioli L, Anderloni A, Fugazza A, Finati E, Pellegatta G, Carrara S, Occhipinti P, Buda A, Fuccio L, Manno M, Hassan C. Novel 1-L polyethylene glycol + ascorbate versus high-volume polyethylene glycol regimen for colonoscopy cleansing: a multicenter, randomized, phase IV study. Gastrointest Endosc. 2021 Oct;94(4):823-831.e9. doi: 10.1016/j.gie.2021.04.020. Epub 2021 Apr 30. PMID 33940043